CLINICAL TRIAL: NCT07198087
Title: A Phase 1, Open-Label, Parallel-Group Study to Investigate the Pharmacokinetics of Tirabrutinib in Participants With Mild, Moderate, and Severe Hepatic Impairment Compared to Healthy Participants
Brief Title: A Study to Investigate the Pharmacokinetics of Tirabrutinib in Participants With Mild, Moderate, and Severe Hepatic Impairment Compared to Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ONO-4059-16
Record Dates: First submitted 2025-08-31; First posted 2025-09-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL)
Keywords: 4059; 4059-16; Tirabrutinib
MeSH Terms: interventions — tirabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tirabrutinib (Mild Hepatic Impairment) (Experimental): Participants received a single dose of Tirabrutinib 80 mg administered orally on Day 1.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib (Moderate Hepatic Impairment) (Experimental): Participants received a single dose of Tirabrutinib 80 mg administered orally on Day 1.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib (Severe Hepatic Impairment) (Experimental): Participants received a single dose of Tirabrutinib 80 mg administered orally on Day 1.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib (Normal Hepatic Function) (Experimental): Participants received a single dose of Tirabrutinib 80 mg administered orally on Day 1.
  Interventions: Drug: Tirabrutinib

INTERVENTIONS:
Drug: Tirabrutinib — Administered orally

SUMMARY:
A study to investigate the pharmacokinetics of tirabrutinib in participants with mild, moderate, and severe hepatic impairment compared to healthy participants

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, age 18 to 75, inclusive, at the time of informed consent.
* BMI between 18 and 40 kg/m2, inclusive, at Screening.
* Continuous non-smokers or smokers who smoke 20 cigarettes or fewer per day.
* Willingness and ability to swallow study intervention tablets.
* Estimated glomerular filtration rate (eGFR) of 45 mL/minute or higher calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) 2021 creatinine equation at Screening.
* Chronic and stable hepatic impairment conforming to Child-Pugh classification A, B, or C, and documented by medical history and a physical examination.
* Adequate bone marrow, renal, and hepatic function at Screening.
* Healthy participants matched to participants with hepatic impairment with regard to sex, BMI (±20%) and age (±10 years), and determined to have no clinically significant deviations from normal in their medical history, physical examination, ECG, and clinical laboratory determinations.

Exclusion Criteria:

* Participant is mentally or legally incapacitated or has significant emotional problems at the time of the Screening visit or such issues can be expected during the conduct of the study.
* History of liver transplant.
* History of any major invasive surgery within 28 days before dosing, or minor invasive surgery within 7 days before dosing.
* Presence of any clinically significant, ongoing systemic bacterial, fungal, or viral infections (including upper respiratory tract infections, but excluding localized cutaneous fungal infections), based on the judgement of the investigator or history of an infection (other than nail trichophytosis) that requires hospitalization or an intravenous antibiotic within 28 days before dosing.
* History or suspicion of interstitial lung disease.
* History of stroke or intracranial hemorrhage within 6 months before dosing.
* History of bleeding diathesis (eg, hemophilia, von Willebrand disease).
* History of Stevens-Johnson syndrome or toxic epidermal necrolysis.
* In the opinion of the investigator, any clinically significant condition that may affect tirabrutinib absorption, including gastric restrictions and bariatric surgery (eg, gastric bypass). Participants with cholecystectomy will be allowed to participate.
* Positive results at Screening for human immunodeficiency virus (HIV).
* History of hypersensitivity or anaphylaxis to tirabrutinib.
* In the opinion of the investigator, participant has been on a diet incompatible with the on-study diet within 28 days before dosing.
* Donation of blood >500 mL or significant blood loss within 56 days before dosing.
* Plasma donation within 7 days before dosing.
* Is working at or has an immediate family member (spouse or children) who works at the study site or is a staff member of the sponsor and directly involved in this trial.
* Dosed in another clinical trial within 28 days or within a period equivalent to 5 half-lives of the investigational drug (whichever is longer) before dosing.
* Have QT interval corrected according to Fridericia's formula (QTcF) >450 ms or deemed clinically abnormal by the investigator at Screening.
* Intake of grapefruit, Seville orange, or herbal preparations containing St. John's Wort within 14 days before dosing.
* Engagement in strenuous exercise (eg, moving large bulky items, bodybuilding) within 14 days before dosing.
* Receipt of any medication (including prescription or over-the-counter medicines, vitamin supplements, natural or herbal supplements) within 14 days before dosing.
* Receipt of any CYP3A4 inducers, P-glycoprotein inducers, or strong CYP3A4 inhibitors within 14 days before dosing.
* Have hepatic encephalopathy of Grade 2 or above at Screening.
* History or presence of drug abuse within 6 months before dosing.
* ALT or AST ≥ 3 × upper limit of normal (ULN) on clinical laboratory tests at Screening. Participants with ALT or AST values ≥2 × ULN and <3 × ULN may be enrolled at the discretion of the investigator following consultation with the medical monitor. Acknowledging the medical state of the population enrolled, participants with hepatitis B and C are not specifically excluded.
* History or presence of alcoholism and/or drug abuse within 6 months before dosing. Alcohol abuse is defined as 8 or more drinks per week for a woman or 15 or more drinks per week for a man.
* Systolic blood pressure (BP) < 90 mm Hg or > 150 mm Hg and/or diastolic BP < 40 mm Hg or > 95 mm Hg sustained for > 5 minutes while resting in a seated position at Screening.
* Seated pulse rate is < 40 beats per minute (bpm) or > 99 bpm at Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of tirabrutinib: Cmax | 72 hour
Pharmacokinetic parameter of tirabrutinib: Tmax | 72 hour
Pharmacokinetic parameter of tirabrutinib: AUClast | 72 hour
Pharmacokinetic parameter of tirabrutinib: AUCinf | 72 hour
Pharmacokinetic parameter of tirabrutinib: T1/2 | 72 hour
Pharmacokinetic parameter of tirabrutinib: CL/F | 72 hour
Pharmacokinetic parameter of tirabrutinib: Volume of distribution (Vd) | 72 hour
Protein binding ratio of tirabrutinib in plasma | 72 hour

SECONDARY OUTCOMES:
Safety and tolerability: Vital signs (pulse rate) | 72 hour
Safety and tolerability: Vital signs (blood pressure) | 72 hour
Safety and tolerability: Vital signs (respiratory rate) | 72 hour
Safety and tolerability: Vital signs (body temperature) | 72 hour
Safety and tolerability: Number of participants with clinically significant abnormal 12-lead electrocardiogram (ECG) parameters (RR, PR, QRS, QT, QTcF) | 72 hour
  The number of participants with clinically significant abnormal values in any of the following ECG parameters will be reported: RR, PR, QRS, QT intervals, and QTcF.
Safety and tolerability: Number of participants with clinically significant abnormal laboratory values | 72 hour
  The number of participants with clinically significant changes in any laboratory value (hematology, clinical chemistry, coagulation, and urinalysis) will be reported.
Safety and tolerability: Adverse events (AEs) | 72 hour

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (2):
- United States (2):
  - Panax Clinical Research, Miami Lakes, Florida
  - Orlando Clinical Research Center, Inc., Orlando, Florida

IPD SHARING:
Plan to Share IPD: No